CLINICAL TRIAL: NCT06347406
Title: Effects of Combined Physiotherapy Management and Education on Physiological Functions and Quality of Life Among Individuals With Patellofemoral Pain
Brief Title: Effects of Combined Physiotherapy Management and Education
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fakulti Sains Kesihatan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FSKesihatan
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Physical Therapy Modalities; Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood flow restriction combined with physiotherapy and education (Experimental): Blood flow restriction, combined with physiotherapy exercises and patient education
  Interventions: Other: Blood flow restriction combined with physiotherapy and education
- Control Group (Placebo Comparator): physiotherapy exercises
  Interventions: Other: Blood flow restriction combined with physiotherapy and education

INTERVENTIONS:
Other: Blood flow restriction combined with physiotherapy and education — Blood flow restriction Physiotherapy exercises Education
  Other Names: Linda Physiotherapy programme

SUMMARY:
This observational study aims to determine the effects of combined physiotherapy programs and education in patellofemoral pain syndrome. The main questions it aims to answer are:

* Are there any effects of combined physiotherapy program among individuals with PFPS on:

  i) Pain ii) Muscle functions (strength, muscle bulk, flexibility) iii) Knee muscle functional performance (anteromedial lunge, step-down, bilateral squat, and balance and reach) iv) Kinesiophobia v) Quality of life Participants will be
* Measure for the anthropometrics data including body weight, height, and BMI.
* Answer the Numerical Pain Rating scale
* Abswe Malay version of KOOS-PF and TAMPA scale.
* Once they finished with the questionnaire, the participants will be stationed into station 1 (HDD), station 2 (Realtime Ultrasound) and station 3 (Dartfish Motion Analysis) Treatment they will receive
* Blood flow restrictions cuff with physiotherapy exercises
* Patient education Researcher will compare Blood flow exercises combined with physiotherapy exercises and education (Group A) with Physiotherapy exercises (Group B) to see if there is an effect on i) Pain ii) Muscle Functions (strength, muscle bulk, flexibility iii) Functional performance (anteromedial lunge, step-down, bilateral squat, balance, and reach) iv) Kinesiophobia v) Quality of life

DETAILED DESCRIPTION:
The participants who volunteered will be screened for inclusion and exclusion criteria. Prior to the assessments and examinations, the physiotherapist in charge will explain the study and will get consent from the participants. This study will follow the Consort RCT 2010 guidelines.

Then the participants will go into randomization sequence before they go into the interventions. The participants will go into block randomization. The participants will be blocks into color (Blue for Experimental group, Red for control group). This study will be double blinded. The blinded person will be the accessors and the participants.

Then they will complete the demographic questionnaire which will include questions on personal data, health status, medical illness, past medical history, simple questions on their pain, site of pain with the assistance by the researchers to read the questions as most of the participants is illiterate.

Then the participants will be measure for the anthropometric data including body weight, height and BMI.

The participants will answer the Numerical Pain Rating scale, KOOS-PF Malay version and TAMPA scale. Then they will proceed with station 1 (HHD which measure strength), station 2 (Real time ultrasound which measure muscle bulk) and then station 3 (Dartfish motion analysis for knee functional performance test (anteromedial lunge, step-down, single-leg press, bilateral squat, and balance and reach) using the Dartfish software.

Station 1 (HDD) will be conducted by a physiotherapist who specially trained to do the HDD. The physiotherapist will then measure the Quadriceps and Hamstrings. These were the procedures that the physiotherapist needs to do:

1. Quadriceps Procedure: Allow for free hanging of the leg at a 90-degree angle. Place the HDD just proximal to the lateral and medial maleolis. Instruct the individual to reach full knee extension effort in 1-2 seconds and then sustain it for an additional 2-3 seconds. Ascertain that the subject's leg is fully stretched away from their body.
2. Hamstrings Procedure: In a prone position, the knee was flexed to 15° and 90° of flexion, as determined by ocular judgement. The examiner positioned the HHD at the subject's heel and gradually increased the force applied to the calcaneal for 1-2 seconds. The individual will be instructed to resist the applied force.In a prone position, the knee was flexed to 15° and 90° of flexion, as determined by ocular judgement. The examiner positioned the HHD at the subject's heel and gradually increased the force applied to the calcaneal for 1-2 seconds. The individual will be instructed to resist the applied force. In a prone position, the knee was flexed to 15° and 90° of flexion, as determined by ocular judgement. The examiner positioned the HHD at the subject's heel and gradually increased the force applied to the calcaneal for 1-2 seconds. The individual will be instructed to resist the applied force.

After the participant completed with the station 1, then he/she will be proceeded with Station 2 (Real time ultrasound).

Procedure: To prevent hip external rotation when supine, a strap was attached around both participant's feet. A 38 mm, 13e18Hz linear transducer was placed above each pen-marked spot to get ultrasonic readings (HDI3000 by Advanced Technology Laboratories, California). The photographs were taken by a technician or a physiotherapist (which one is available) who had received training in real-time ultrasonography. Gain was increased until muscle borders appeared on the screen, and the picture depth was adjusted until the femur was visible in the screen's central. Each muscle, namely the vastus medialis (VM), the vastus lateralis (VL), the vastus intermedius (VI), the rectus femoris (RF), and the vastus medialis (VM), semimembranousus (SM), semitendinosus (ST) and Biceps Femoris (BF). Iliotibial band (ITB), tenssofacialate (TFL) and gastrocnemius (GSN) will be photographed three times. To minimize muscular stiffness, the transducer head was adequately covered in ultrasonic gel.

Once completed with the station 2, then the participant will proceed with station 3 (Knee Muscle performance Test with Dartfish motion software). This station will be conducted by a physiotherapist who trained in Dartfish motion analysis software.

Procedure:

The participant is dressed in compression shorts and shirt that fit tightly to the body. The lower extremity model that utilizes four markers placed in various locations from the acromion joint, greater trochanteric, medial tuberosity of femur down to the lateral malleolus. After the marker is install on the participant body, they are requiring to perform these movements:

Anteromedial lunge left and right: The subject is positioned behind a starting line. The subject lunges forward with the uninvolved limb so that the front leg bends to 90 degrees and crosses the midline. The patient must keep his or her balance and maintain an upright trunk posture. The participant is then instructed to perform as many lunges in 30 seconds; lunges that do not meet the 80% level are not recorded. The lunge is not included in the count if the subject deviates from the path of motion or takes an extra step.

Step-down, left and right: The step-down is a unilateral test done from an 8-inch (20.32-centimeter) high platform. Participant take a step forward and lower themselves to the ground. Only the heel of the down leg brushes the floor before returning to full knee extension. This is considered one repeat. This to allow to calculate the time take to complete one cycle and speed (Refer to Appendix E). The trunk, hip, knee and ankle ROM is calculate when the both foot touches the step and when the test foot starting to go down to the ground. Both limbs are put to the test

Bilateral squat: The participant begin by standing with their legs fully extended, shoulders shoulder-width apart, and their weight evenly distributed on both limbs. Participant lower their bodies to a 90 degrees knee position before returning to full extension. A complete cycle of straight standing to 90 degrees of knee flexion and back to straight standing constitutes one repeat (speed and time of this cycle will be calculate.

Balance and reach (to measure distance) : Behind a start line, the subject begins the test. The participant extends one leg straight forward until the heel contacts the floor, with the rear (test) leg bearing most of the body weight. The unaffected limb is put to the test first. Measurement between the starting point to end point will be calculated

Once they completed the questionnaire and assessment, then the participant will proceed with the interventions.

The participant will need to strap proximal parts of the lower limb with 40% of subject's RECOVER FUN AIR CUFF WITH PUMP. The timer will be set up to 10 minutes during the intervention for the participants' to release the pressure of the cuff. The participants' will rest on the chair for 5 minutes. The participants will need to perform physiotherapy exercises with the cuff on.

Education booklet will be designed to educate the participants about the PFPS, advice and importance of exercises.

The contain of this booklet consist of:

1. What is PFPS
2. What causes PFPS
3. What are the symptoms of PFPS?
4. Pain gate theory
5. Importance of treatment
6. Exercises
7. Frequently asked questions

Follow up Participants will need to come in for intervention for three times a week for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Pain and disability in at least three of the following activities involving pain around the patella
2. Scored in KOOS-PF

Exclusion Criteria:

1. Failure to regularly continue treatment sessions
2. A history of knee surgery and severe trauma with meniscus or ligament tear within 6 months
3. Went for acupuncture treatment
4. Undergone any type of surgical procedure
5. Pregnancy, cancer, secondary osteoarthritis and various rheumatologic diseases, and symptoms of abnormal neurological examination of sensation, movement, and reflexes

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating | 4 months
  On a Numerical Pain Rating Scale, often known as an NPRS, patients are asked to circle the number between 0 and 10, 0 and 20, or 0 and 100 that most properly portrays the intensity of pain that they are experiencing
The Knee injury and Osteoarthritis Outcome Score for patellofemoral pain and osteoarthritis (KOOS-PF) | 4 months
  The KOOS-PF subscale is used to assess pain and function in the patellofemoral joint. The 11-point KOOS-PF, which was created in collaboration with healthcare professionals, demonstrated adequate measuring qualities and is recommended for clinical and research usage in patients suffering from patellofemoral pain
Tampa Scale | 4 months
  The Tampa Kinesiophobia Scale (TSK) is a self-assessment measure used to determine a person's fear of movement-related pain who suffers from musculoskeletal discomfort
Hand held dynamometer (HDD) | 4 months
  The examiner holds a small portable gadget against the patient's limb during a maximal isometric contraction. The equipment can test both the proximal and distal muscles of all extremitie
Knee Muscle performance Test with Dartfish software | 4 months
  Dartfish data will be used to process the action of anteromedial lunge, step-down, bilateral squat, and balance and reach during simultaneous digital video acquisition. In other words, Dartfish programme will generate data. All of these movements will be measured with Dartfish software
Real time ultrasounds | 4 months
  The thickness and length of the superficial quadriceps muscles (VMO, VL, VL, and RF).

CONTACTS AND LOCATIONS:
Locations (1):
- Fakulti Sains Kesihatan, Shah Alam, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No